CLINICAL TRIAL: NCT06577064
Title: Sacral Erector Spinae Block for Pilonidal Sinus Surgery: A Randomized Controlled Trial
Brief Title: Sacral Erector Spinae Block for Pilonidal Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, rabab Mohammad habeeb, Principal investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANET6_2
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: andomized controlled trial.
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacral erector spinae plane block Group (Active Comparator): 30 ml of 0.2% ropivacaine will be injected in the plane between the ESM and sacrum on each side While the patient is in prone position
  Interventions: Procedure: Sacral erector spinae plane block
- non-intervention group (Placebo Comparator): patients will receive general anesthesia plus scheduled analgesia protocol in the form of morphine sulphate I.V. 1 mg every 5 minutes if NRS more than 5 till maximum dose 10 mg
  Interventions: Procedure: Sacral erector spinae plane block

INTERVENTIONS:
Procedure: Sacral erector spinae plane block — 30 ml of 0.2% ropivacaine will be injected in the plane between the ESM and sacrum on each side

SUMMARY:
The incidence of pilonidal sinus disease (PD) is estimated to be around 26/100,000 individuals mostly men.PD can cause the development of abscess or a draining sinus tract and that may lead to a loss of productive power and long-term morbidity.Different surgical technique approaches were proposed for treatment with different rates of success.

DETAILED DESCRIPTION:
Sacral erector spinae plane block was first described by Tulgar et al. To provide sensory blockade in the parasacral region in two cases who had pilonidal sinus surgeries. Since then, the block was used for multiple surgeries like anorecatal, hip surgery and parasacral reconstructive surgeries.After obtaining the ethical committee approval from Menoufia University. patients scheduled for pilonidal sinus surgery will be randomly allocated into one of two groups Patients will be randomized to a study group using a computer-generated random number table, and the allocation concealment will be performed using a sealed envelope technique.The sealed opaque envelopes will be kept locked in dedicated research safe and will be accessed by a research coordinator only when a patient consented for the study. The anesthetist will perform the intervention with the doses and concentration of drugs as per the protocol.

The patients and the follow up researcher will be blinded to the type of intervention used. The patient follow-up time will be scheduled intraoperatively PACU, 1 hour and 24hours postoperatively. The anesthetist who did the intervention will have no access to the reported documents or contact with the patient postoperatively.

For induction of anesthesia all patients will receive medication as per the facility protocol where propofol 1-2mg/Kg, fentanyl 2μg/Kg (actual BW), rocuronium 0.5 mg/kg will be used for induction and an endotracheal tube intubation will be inserted to secure the airway. After intubation and confirmation of endotracheal tube placement by auscultation and capnography, the patient will be turned into prone position.

Maintenance of anesthesia will be maintained by sevoflurane 1-1.2 MAC and rocuronium 0.1mg/kg guided by the TOF. All patients will receive multimodal analgesia in the form of paracetamol 1gm and parecoxib 40 mg (Pizer manufacturing Belgium). After exclusion of other causes of tachycardia and hypertension Morphine 2mg increments will be administrated to keep the heart rate or blood pressure within 20 percent of the patient's baseline parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* ASA physical status 1-3

Exclusion Criteria:

1. ASA >3
2. Opioid use within the previous 3 months
3. Deranged coagulation parameters
4. Patient refusal
5. Allergy to local anesthetic medication.
6. Preoperative neurological deficits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Pain score | 24 hours
  NRS scor for post operative pain scale from 0 to 100

SECONDARY OUTCOMES:
Opioid consumption. | 24 hours
  Total opioid consumbtion in mg
Lower limb motor affection | 24 hours
  Modified Bromage scale for motor affection from 1 to 6
Adverse effects | 24 hours
  Side effect as nausea, vomiting, itching will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: rabab M habeeb, Principal Investigator — Menoufia University
Locations (1):
- Faculty of Medicine Menoufia University, Cairo, Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No